CLINICAL TRIAL: NCT02410382
Title: A Phase II Randomized Study of Short-Term Dexamethasone Versus Placebo for Fatigue in Patients Receiving Radiation Alone or Radiation and Chemotherapy for the Treatment of Head and Neck and Non-Small Cell Lung Cancers
Brief Title: Dexamethasone for Treatment of Radiation-related Fatigue in Patients Receiving RT for Head-neck and Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: IRB suspension, did not resume
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1408439554
Record Dates: First submitted 2015-03-30; First posted 2015-04-07 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-04

CONDITIONS: Head and Neck Cancer; Non-small Cell Lung Cancer
Keywords: cancer; radiation therapy; chemotherapy; dexamethasone; corticosteroids
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Dexamethasone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 Placebo (Placebo Comparator): Subjects receiving radiation therapy or radiation and chemotherapy randomly assigned to placebo bid for 14 days
  Interventions: Drug: Placebo
- Arm 2 Dexamethasone (Active Comparator): Subjects receiving radiation therapy or radiation and chemotherapy randomly assigned to dexamethasone 4 mg bid for 14 days
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — oral dexamethasone 4 mg bid for 14 days
  Other Names: corticosteroid
  Arms: Arm 2 Dexamethasone
Drug: Placebo — oral placebo
  Arms: Arm 1 Placebo

SUMMARY:
This study will look at how dexamethasone and placebo influence radiation fatigue, quality of life and number of treatment days missed during radiation therapy or radiation therapy and chemotherapy for cancer.

DETAILED DESCRIPTION:
Subjects will randomly receive either dexamethasone or placebo and begin the study medication during the midpoint of their radiation treatment. Study medication will be taken for 14 straight days then stopped. Fatigue and quality of life will be measured weekly with short patient completed surveys. The number of breaks taken during radiation treatment will also be tracked. For safety, blood sugar levels will be checked with finger stick blood draws because dexamethasone is known to cause these levels to increase. Study participation will be approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* confirmation of head & neck cancer (stage I-IV) or non-small cell lung cancer (stage II & III)
* Undergoing treatment with either radiation alone or in combination with chemotherapy
* Normal cognition and willingness to complete fatigue and quality of life forms, patient observation form, and pill diary

Exclusion Criteria:

* Hypersensitivity to dexamethasone or corticosteroids or Equal sugar substitute
* Corticosteroid within the past 30 days prior to study enrollment for greater than one week duration
* Planned Stereotactic Body Radiation Therapy (SBRT)
* Active psychosis
* Current pregnancy
* Active peptic ulcer disease or evidence of gastrointestinal bleed
* Current active tuberculosis or systemic fungal infection
* Previous diagnosis of diabetes mellitus
* Acute febrile illness
* Known human immunodeficiency virus or acquired immunodeficiency syndrome
* Major surgery within two weeks of study enrollment of which the patient has not recovered
* Psychostimulant use in the past 30 days prior to registration
* History of phenylketonuria (PKU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2014-08-27 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sun Yi, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study was terminated and data coordinator is no longer in the institution. Sincere efforts were made to gather and report the data, however, no data are available since the study records cannot be located.
Groups:
- Arm 2 Dexamethesone: Subjects receiving radiation therapy or radiation and chemotherapy randomly assigned to dexamethasone 4 mg bid for 14 days
  Dexamethasone: oral dexamethasone 4 mg bid for 14 days
Period: Overall Study
Arm/Group | Arm 1 Placebo | Arm 2 Dexamethesone
Started | 0 | 0
Completed | 0 (Study was terminated by IRB - attempts made to obtain info were unsuccessful.) | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated by IRB - attempts made to obtain info were unsuccessful.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 Placebo | Arm 2 Dexamethesone | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Fatigue Measured by FACIT-F Version 4 Fatigue Score
Description: To compare the effects of dexamethasone and placebo on radiation fatigue using validated measures
Time Frame: 12 weeks
Population: Data were collected but could not be analyzed. Study terminated by IRB and any data that were gathered, are lost. No data are available for this assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 Placebo | Arm 2 Dexamethesone
Number analyzed (Participants) | 0 | 76
Participants | 0 | 0

2. Secondary Outcome: Quality of Life as Measured by FACIT-F Version 4 Well-Being Score
Description: To determine the effect of dexamethasone on QoL and radiation therapy treatment interruption
Time Frame: 12 weeks
Population: as for outcome 1
Arm/Group | Arm 1 Placebo | Arm 2 Dexamethesone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Data unavailable; study terminated. Good faith attempts made to locate any data have been unsuccessful.
Description: Data unavailable; study terminated. Good faith attempts made to locate any data have been unsuccessful.
Arm/Group | Arm 1 Placebo | Arm 2 Dexamethesone
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT02410382/Prot_SAP_000.pdf